CLINICAL TRIAL: NCT04685590
Title: Phase II Clinical Trial to Evaluate the Safety and Feasibility of Senolytic Therapy in Alzheimer's Disease
Brief Title: Senolytic Therapy to Modulate the Progression of Alzheimer's Disease (SToMP-AD) Study
Acronym: SToMP-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00067429
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease, Early Onset; Mild Cognitive Impairment
Keywords: amnestic mild cognitive impairment; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Dasatinib (D) is given as (1) 100mg capsule daily for 2 consecutive days (Sprycel®, Bristol Myers Squibb). Quercetin (Q) will be given as (4) 250 mg capsules daily (total 1000 mg daily) for the same 2 consecutive days (Thorne Research). Both are administered orally.
  Interventions: Drug: Dasatinib + Quercetin
- Placebo (Placebo Comparator): Matching placebo capsules following the same administration protocol as the experimental treatment - administered once daily (1st dose of each cycle will be given, supervised, at the clinic visit; the 2nd dose will be taken at home) for 2 consecutive days followed by a 13-day (+/- 2 day) no-drug period for 12 consecutive weeks for 6 rounds of administration.
  Interventions: Other: Placebo Capsules

INTERVENTIONS:
Drug: Dasatinib + Quercetin — D+Q will be administered once daily (1st dose of each cycle will be given, supervised, at the clinic visit; the 2nd dose will be taken at home) for 2 consecutive days followed by a 13-day (+/- 2 day) no-drug period for 12 consecutive weeks for 6 rounds of administration.
  Arms: Treatment
Other: Placebo Capsules — Matching placebo capsules following the same administration protocol as the experimental treatment - administered once daily (1st dose of each cycle will be given, supervised, at the clinic visit; the 2nd dose will be taken at home) for 2 consecutive days followed by a 13-day (+/- 2 day) no-drug period for 12 consecutive weeks for 6 rounds of administration.
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the safety, feasibility, and efficacy of senolytics in older adults with amnestic mild cognitive impairment (MCI) or early-stage AD (Clinical Dementia Rating (CDR)=0.5 or 1) who are tau PET positive

DETAILED DESCRIPTION:
This study is a Phase II multi-site, randomized, double-blind placebo controlled trial to determine safety, feasibility, and efficacy of senolytics in older adults with amnestic mild cognitive impairment (MCI) or early-stage AD (Clinical Dementia Rating (CDR)=0.5 or 1) who are tau PET positive.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 60 years and older at study entry
2. Both sexes
3. All ethnicities
4. Diagnosis of amnestic mild cognitive impairment (aMCI) or early Alzheimer's disease (AD)
5. Elevated tau protein as determined by CSF performed during screening. Evidence of elevated tau from previously available CSF samples will also be allowed for eligibility determination.
6. FDA-approved medications for AD (e.g. donepezil, rivastigmine, galantamine) are permitted as long as the participant has been maintained on a stable dose for at least three months prior to study entry.
7. Labs: Normal blood cell counts, normal liver and renal function without clinically significant excursions as determined by coordinating center Medical Monitor. Total cholesterol <240 mg/dl, HbA1c ≤ 7%.
8. Prothrombin Time (PT)/Partial Thromboplastin Time (PTT)/International Normalized Ratio (INR) within normal limits.
9. Participants must have the ability to provide written consent or be accompanied by a Legally Authorized Representative designated to sign informed consent (if determined not to have decision capacity).
10. Participants must have a study partner who agrees to participate throughout the duration of the study. The study partner must have frequent and sufficient contact (approximately 10 hours per week) with the participant and be able to provide accurate information regarding the participant's cognitive and functional abilities.
11. Participants must have no travel plans that would interfere with scheduling visits following consent over the 12 months of study duration.
12. Must speak English fluently and have at least six years of formal education.
13. Participants must be fully vaccinated against COVID-19 with the primary vaccine series per CDC recommendations, with any dose of the vaccine received at least 30 days prior to initiation of the study drug. COVID boosters are allowed during study intervention period when scheduled at least four days before or after administration of the investigational product.

Exclusion Criteria:

1. Body mass index (BMI)>40 kg/m2.
2. Average QTcF (from 3 ECGs obtained at least one minute apart) at screening of ≥450msec in males and ≥460msec in females.
3. MRI contraindications including claustrophobia, the presence of metal (ferromagnetic) implants, or cardiac pacemaker.
4. Pregnancy or possible pregnancy.
5. Any significant neurologic disease other than prodromal or early AD including Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
6. Current or history of alcohol or substance abuse or dependence within the past 2 years per Diagnostic and Statistical Manual of Mental Disorders (DSM V criteria).
7. Endorsement of current suicidality or suicidal ideation on the screening C-SSRS.
8. Uncontrolled diabetes (HbA1c > 7% or the current use of insulin or sulfonylureas).
9. Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg) based on two or more readings and as determined by the PI/study clinician.
10. eGFR < 10 ml/ min/ 1.73 m2.
11. Myocardial infarction, angina, stroke, or transient ischemic attack in the past 6 months.
12. Chronic heart failure.
13. Presence of significant liver disease with total bilirubin >2X upper limit.
14. Inability to tolerate oral medication.
15. Participants taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4 (e.g., cyclosporine, tacrolimus, or sirolimus).
16. Participants currently taking drugs that induce cellular senescence: alkylating agents, anthracyclines, platins, other chemotherapy.
17. Participants on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.) other than low dose aspirin unless able to be held for 2 days prior to LP and with the documented approval of the prescribing clinician.
18. Participants taking H2 antagonists or proton pump inhibitors who are unable or unwilling to reduce or hold therapy for at least 2 days prior to and during each of the 2-day courses of Dasatinib plus quercetin dosing. Instead, subjects may use antacids prior to and during each of the 2-day courses of Dasatinib plus quercetin dosing.
19. Concomitant use of strong CYP3A4 inhibitors.
20. Co-enrollment in another ADRD research study with a potentially disease-modifying intervention or study drug that may impact senescent cells. Participants previously enrolled in a study meeting these criteria are eligible to screen after a washout period of ≥6 months from date of last dose to date of screening.
21. Presence of any condition that the Investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial.
22. Use of anti-amyloid therapies (e.g. aducanumab, lecanamab).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) and Adverse Events (AEs) in treatment group as compared to placebo group | Baseline to Week 48
  Adverse Events (AEs) and SAEs will be collected at each in-person visit and at scheduled telephone visits from baseline to week 48. Incidence of SAEs between groups (treatment vs. placebo) will be reviewed by the Data Safety Monitoring Board (DSMB) for clinical significance.

SECONDARY OUTCOMES:
Change in cellular senescence blood marker Senescence-Associated Secretory Phenotype (SASP) composite score | Baseline to Week 12
  Composite score (average z-score of log-transformed values) of ten primary SASP factors measured in blood.
Change in cellular senescence blood marker Cluster of Differentiation 3 (CD3) in blood | Baseline to Week 12
  Primary markers of cellular senescence CD3 measured in blood.
Change in cellular senescence blood marker cyclin-dependent kinase inhibitor 2A (p16INK4A+) in blood | Baseline to Week 12
  Primary markers of cellular senescence p16INK4A+ measured in blood.
Change in cellular senescence blood marker T cells in blood | Baseline to Week 12
  Primary markers of cellular senescence T cells measured in blood.
Change in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) slope | Baseline to Week 48
  CDR is calculated on the basis of testing six different cognitive and behavioral domains such as memory, orientation, judgment and problem solving, community affairs, home and hobbies performance, and personal care. The CDR is based on a scale of 0-3: no dementia (CDR = 0), questionable dementia (CDR = 0.5), MCI (CDR = 1), moderate cognitive impairment (CDR = 2), and severe cognitive impairment (CDR = 3). The six domains are often summed to create a 0 - 18 "sum of the boxes" score. CDR-SB has been shown to demonstrate sensitivity to cognitive changes associated with progression of amnestic mild cognitive impairment (aMCI) and early Alzheimer's Disease (AD).
Change in the 14 - item Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog 14) slope | Baseline to Week 48
  A psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates more impairment. Scores from the original portion of the test range from 0 (best) to 65 (worse), and are added to the mean of the words not immediately recalled (max of 10) and the number of items not recalled after a delay (ranging from 0-10) all total the maximum score of 85. A positive change indicates cognitive worsening.
Change in Positron Emission Tomography (PET) - Computed Tomography (CT) - brain tau pathology | Baseline to Week 48
  Tau levels in the brain will measured by 18F AV1451 PET imaging to assess target engagement of dasatinib and quercetin (D+Q) and impact on brain tau as a relevant Alzheimer's Disease (AD) biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Orr, PhD, Principal Investigator — Washington University School of Medicine
Locations (5):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States
- Spain (4):
  - Fundación ACE Clinical Site, Barcelona
  - Hospital Clínic de Barcelona Site, Barcelona
  - Sant Pau Clinical Site, Barcelona
  - FISEVI Clinical Site, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzales MM, Krishnamurthy S, Garbarino V, Daeihagh AS, Gillispie GJ, Deep G, Craft S, Orr ME. A geroscience motivated approach to treat Alzheimer's disease: Senolytics move to clinical trials. Mech Ageing Dev. 2021 Dec;200:111589. doi: 10.1016/j.mad.2021.111589. Epub 2021 Oct 21. PMID 34687726
- [Derived] Guerrero A, De Strooper B, Arancibia-Carcamo IL. Cellular senescence at the crossroads of inflammation and Alzheimer's disease. Trends Neurosci. 2021 Sep;44(9):714-727. doi: 10.1016/j.tins.2021.06.007. Epub 2021 Aug 5. PMID 34366147